CLINICAL TRIAL: NCT01356693
Title: Randomized,Double-blind, Placebo Controlled Clinical Trial to Evaluate the Efficacy of the Phytotherapic Compound "Bromelin" on Acute Irritative Cough
Brief Title: Bromelin, a Compound Prepared With Ananas Comocus Extract and Honey, for Acute Cough
Acronym: BROMETOSS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Emanuel Sávio Cavalcanti Sarinho, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Brom1
Record Dates: First submitted 2011-05-12; First posted 2011-05-19 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-03

CONDITIONS: Cough, Acute
Keywords: Cough; Common cold; Child; Adolescent
MeSH Terms: conditions — Cough; Common Cold | interventions — Bromelains

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Experimental): Bromelin. Extract from Ananas comosus, 3,3g on vehicle (methylparaben, propylparaben, honey from apis mellifera, sodium benzoate, ethylic alcohol, water) 5ml.
  Interventions: Drug: Bromelin
- Placebo (Placebo Comparator): Placebo comparator with the same characteristics of experimental drug, 5ml, single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bromelin — Ananas comosus extract (3,3g) on vehicle: methylparaben, propylparaben, honey from Apis mellifera, sodium benzoate, ethilic alcohol, water) 5ml. Given in single dose.
  Other Names: Bromelein; Ananas comosus extract
  Arms: Active drug
Drug: Placebo — Placebo with mimicking characteristics of experimental drug
  Arms: Placebo

SUMMARY:
Cough is the most bothersome symptom for patients with the common cold.

The objective of the study is to compare the phytotherapic "Bromelin", a compound preparation of honey from the bee apis mellifera with the extract of the pineapple (Ananas comosus) with placebo in reducing cough episodes in patients with the common cold.

DETAILED DESCRIPTION:
Common cold is very frequent and cough is one of the most troublesome symptoms. Over-the-counter medications are used by patients without prescription, many times with important side effects.

Bromelin, a compound made with honey and pineapple extract could offer cough symptomatic relief as a soothing agent.

This study aims to compare this compound with placebo in reducing cough in patients with common cold in an clinical trial designed in conformity to CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* cough for less than 24 hours
* common cold symptoms : nasal obstruction, headache, myalgias, runny nose.

Exclusion Criteria:

* declared chronic pulmonary diseases declared Nervous diseases declared Diabetes declared cardiac diseases known primary or secondary immunodeficiencies

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-11 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change in score in a cough evaluation questionnaire | before and 10 and 30 minutes after the dosing
  A cough score based on number of coughing episodes and subjective 5 item cough score : no cough, mild, moderate, severe, very severe.

SECONDARY OUTCOMES:
Change in Occurrence of gastric symptoms | 10 and 30 minutes
  Question "YES" as answer to questions about gastric symptoms as nausea and/or vomiting after medication

CONTACTS AND LOCATIONS:
Overall Officials: Decio M Peixoto, MD, PhD, Study Director — UFPE; Emanuel SC Sarinho, MD, PhD, Principal Investigator — UFPE
Locations (1):
- Hospital das Clínicas/UFPE, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Smith SM, Schroeder K, Fahey T. Over-the-counter medications for acute cough in children and adults in ambulatory settings. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD001831. doi: 10.1002/14651858.CD001831.pub3. PMID 18253996
- [Background] Widdicombe J, Morice A. Over the counter cough medicines for acute cough. Good quality research is needed. BMJ. 2002 May 11;324(7346):1158. No abstract available. PMID 12008729
- [Background] Gardner JF. Regulation of the threonine operon: tandem threonine and isoleucine codons in the control region and translational control of transcription termination. Proc Natl Acad Sci U S A. 1979 Apr;76(4):1706-10. doi: 10.1073/pnas.76.4.1706. PMID 287010
- [Derived] Peixoto DM, Rizzo JA, Schor D, Silva AR, Oliveira DC, Sole D, Sarinho E. Use of honey associated with Ananas comosus (Bromelin) in the treatment of acute irritative cough. Rev Paul Pediatr. 2016 Dec;34(4):412-417. doi: 10.1016/j.rpped.2016.03.006. Epub 2016 Apr 16. PMID 27181342